CLINICAL TRIAL: NCT05161962
Title: Investigation of the Effect of Oral Care Given by Two Different Methods in Patients Connected to Mechanical Ventilators on the Development of Ventilator-AssociatedPneumonia
Brief Title: Oral Care to Prevent Ventilator-associated Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ASENA KÖSE, research assistant, Ataturk University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AtaturkU-001
Record Dates: First submitted 2021-12-05; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Oral Hygiene, Oral Health; Ventilators, Mechanical
Keywords: Mechanical ventilation; nursing; oral care; pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One group received standard oral care. (Experimental)
  Interventions: Combination Product: One group received standard oral care.; Combination Product: It was applied to the other group by aspiration.
- It was applied to the other group by aspiration. (Placebo Comparator)
  Interventions: Combination Product: One group received standard oral care.; Combination Product: It was applied to the other group by aspiration.

INTERVENTIONS:
Combination Product: One group received standard oral care. — the effect of oral care given by two different methods on the development of ventilator-associated pneumonia in patients connected to mechanical ventilators.
Combination Product: It was applied to the other group by aspiration. — the effect of oral care given by two different methods on the development of ventilator-associated pneumonia in patients connected to mechanical ventilators.

SUMMARY:
This study was conducted to investigate the effect of oral care given by two different methods on the development of ventilator-associated pneumonia in patients connected to mechanical ventilators.

DETAILED DESCRIPTION:
The universe of this research, which was designed as a semi-experimental study, is composed of patients connected to the mechanical ventilator lying in Atatürk University Training and Research Hospital Anesthesia and Reanimation Intensive Care Unit between September 2019 and February 2020. A total of 57 patients, 29 method-1, 28 method-2 groups, met the inclusion criteria of the study. In the data collection phase, 'Patient Identifier Information Form', 'Patient Monitoring Form', 'Oral Assessment Scale' and 'Tracheal Aspirate Culture Result Form' were used. In the evaluation of the data, number and percentage distributions, Kruskal Wallis, Mann Withney-U, Wilcoxon Analysis, Chi-Square test were used.

ELIGIBILITY:
Inclusion Criteria:• Patients on mechanical ventilator who have been in intensive care for at least 48 hours

* Male and female patients over the age of 18
* Patients without thrombocytopenia, leukopenia and oral stomatitis, aphthae, candiasis, gingivitis
* Patients whose respiratory support is provided by a mechanical ventilator
* Patients who are considered to be able to provide mechanical ventilator support for 7 days
* Patients without any respiratory-related infectious pathogens
* Obtaining informed consent from the patient if he/she can give consent or from his/her guardian if he/she is unable to give consent.
* It was determined as patients who did not undergo any intraoral surgical intervention.

Exclusion Criteria: patients with pneumonia Patients younger than 18 years

-

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
oral care application with standard oral care stick | 1 in 6 hours
  Administered with chlorhexidine gluconate solution.
Oral care application with a sucking oral care stick | 1 in 6 hours
  Administered with chlorhexidine gluconate solution.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)